CLINICAL TRIAL: NCT04987307
Title: A Phase 2, Dose-finding, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Safety and Efficacy of Efavaleukin Alfa Induction Therapy in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: Safety and Efficacy of Efavaleukin Alfa in Participants With Moderately to Severely Active Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to meeting a prespecified futility rule and not related to any safety concerns.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20170104; 2021-002537-41 (EudraCT Number)
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; UC; Efavaleukin Alfa
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Efavaleukin alfa (Experimental): Efavaleukin alfa Dose 1 administered by SC injection once every two weeks (Q2W)
  Interventions: Drug: Efavaleukin alfa
- Arm B: Efavaleukin alfa (Experimental): Efavaleukin alfa Dose 2 administered by SC injection Q2W
  Interventions: Drug: Efavaleukin alfa
- Arm C: Efavaleukin alfa (Experimental): Efavaleukin alfa Dose 3 administered by SC injection Q2W
  Interventions: Drug: Efavaleukin alfa
- Arm D: Placebo (Placebo Comparator): Placebo Q2W
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efavaleukin alfa — Efavaleukin alfa will be administered by subcutaneous (SC) injection.
  Other Names: AMG 592
  Arms: Arm A: Efavaleukin alfa; Arm B: Efavaleukin alfa; Arm C: Efavaleukin alfa
Drug: Placebo — Placebo will be administered by SC injection.
  Arms: Arm D: Placebo

SUMMARY:
The main purpose of this study is to evaluate the effect of efavaleukin alfa on induction of clinical remission in participants with moderately to severely active ulcerative colitis (UC).

Participants will be randomized to receive 1 of 3 efavaleukin alfa doses or placebo during a 12-week induction period. Participants who complete the 12-week induction period will have the option to enter an exploratory long-term treatment period for up to 40 weeks (total of up to 52 weeks of treatment) if, in the opinion of the investigator, they may benefit from continued treatment. During the long-term period, participants randomized to efavaleukin alfa will remain on the same efavaleukin alfa blinded dose; participants randomized to placebo who achieved clinical response at week 12 will remain on placebo; and placebo non-responders (ie, participants randomized to placebo who did not achieve clinical response at week 12) will receive efavaleukin alfa in a blinded manner during continued treatment. All participants will complete a safety follow-up visit 6 weeks after their last dose of investigational product.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study specific activities or procedures.
* Men and women aged ≥ 18 to < 80 years at screening visit (≥ 19 to < 80 in South Korea).
* Diagnosis of UC established ≥ 3 months prior to enrollment by clinical and endoscopic evidence and corroborated by a histopathology report. If a histopathology report is not available at screening, then additional biopsies may be taken during the screening period for local histopathology analysis to corroborate.
* Moderately to severely active UC as defined by a modified Mayo score of 5 to 9, with a centrally read endoscopy subscore ≥ 2.
* Has documentation of:

  * A surveillance colonoscopy (performed according to local standard) within 12 months of day 1 visit for participants with pancolitis of > 8 years duration, or participants with left-sided colitis of > 12 years duration, or participants with primary sclerosing cholangitis.
  * At the discretion of the investigator, a colonoscopy (instead of a rectosigmoidoscopy) may be performed as the screening endoscopy for this study.
  * For all other participants, up-to-date colorectal cancer surveillance (performed according to local standard). Participants who do not have a colonoscopy report available in source documentation will have a colonoscopy instead of rectosigmoidoscopy performed as the screening endoscopy for the study.
* Participants must have demonstrated inadequate response, loss of response, or intolerance to at least 1 conventional therapy, biologic therapy, or targeted small molecule therapy (ie, Janus kinase [JAK]-inhibitor or or S1P modulators), as follows:

  1. Conventional therapy failed participants:

     * Corticosteroids (corticosteroid-refractory colitis, defined as signs and/or symptoms of active UC despite oral prednisone [or equivalent] at doses of at least 30 mg/day for a minimum of 2 weeks; or corticosteroid-dependent colitis, defined as: an inability to reduce corticosteroids below the equivalent of prednisone 10 mg/day within 3 months of starting corticosteroids without a return of signs and/or symptoms of active UC; or a relapse within 3 months of completing a course of corticosteroids).
     * History of intolerance of corticosteroids (including, but not limited to, Cushing's syndrome, osteopenia/ osteoporosis, hyperglycemia, or neuropsychiatric side-effects, including insomnia, associated with corticosteroid treatment).
     * Immunomodulators: signs and/or symptoms of persistently active disease despite at least 3 months treatment with one of the following at locally approved doses: oral azathioprine (eg, ≥ 1.5 mg/kg/day) or 6-mercaptopurine (eg, ≥ 0.75 mg/kg/day), or oral azathioprine or 6-mercatopurine within a therapeutic range as judged by thioguanine metabolite testing, or a combination of a thiopurine and allopurinol within a therapeutic range as judged by thioguanine metabolite testing.
     * History of intolerance to at least 1 immunomodulator (including but not limited to nausea/vomiting, abdominal pain, pancreatitis, liver function test abnormalities, and lymphopenia) and have neither failed nor demonstrated an intolerance to a biological medication (anti-tumor necrosis factor [TNF] antibody, anti-integrin antibody, or interleukin [IL]-12/23 antagonists) that is indicated for the treatment of UC.
  2. Biologic or targeted small molecule therapy failed participants: those who demonstrated inadequate response or loss of response or intolerance to biologic therapy for UC (eg, anti-TNF antibodies or IL-12/23 antagonists, anti-integrin antibodies) or targeted small molecules (eg, JAK inhibitors or S1P modulators). The therapy used to qualify the participant for entry into this category must be approved for the treatment of UC in the country of use, at the time of use. Participants must fulfil one of the following criteria:

     * Inadequate response: signs and symptoms of persistently active disease despite induction treatment at the approved induction dosing that was indicated in the product label at the time of use.
     * Loss of response: recurrence of signs and symptoms of active disease during approved maintenance dosing following prior clinical benefit (discontinuation despite clinical benefit does not quality as having failed or being intolerant to UC biological therapy, JAK inhibitor, or S1P modulators).
     * Intolerance: history of intolerance to infliximab, adalimumab, golimumab, vedolizumab, ustekinumab, tofacitinib or other approved biologicals, JAK inhibitors or S1P modulators (including but not limited to infusion-related event, demyelination, congestive heart failure, or any other drug-related adverse event that led to a reduction in dose or discontinuation of the medication).
* If receiving any of the following therapies, participants must have stable dosage for the specified duration:

  * 5-aminosalicylates (ASAs), stable dosage for ≥ 2 weeks prior to screening endoscopy.
  * Oral corticosteroids: prednisone ≤ 20 mg/day or its equivalent, stable dose for ≥ 2 weeks prior to screening endoscopy.
  * Budesonide: extended release tablets 9 mg/day [budensonide MMX], stable dose for ≥ 2 weeks prior to screening endoscopy.
  * Beclomethasone dipropionate: gastro-resistant prolonged-release tablet 5 mg/day, stable dose for >= 2 weeks prior to screening endoscopy.
  * Conventional immunomodulators: azathioprine, 6-mercaptopurine, methotrexate, stable dosage for ≥ 12 weeks prior to screening endoscopy.

Key Exclusion Criteria:

* Diagnosis of Crohn's disease, inflammatory bowel disease unclassified (indeterminate colitis), microscopic colitis, ischemic colitis, or clinical findings suggestive of Crohn's disease.
* Evidence of toxic megacolon, fulminant colitis, intra-abdominal abscess, or stricture/stenosis within the small bowel or colon.
* Participant has had extensive surgery for UC (for example, subtotal colectomy), or is likely to require surgery for the treatment of UC during the study.
* Currently receiving or had treatment within 12 months prior to screening with T cell depleting agents (eg, antithymocyte globulin, Campath).
* Participant has received any of the following prescribed medication or therapy within the specified time period:

  * Anti TNF antibodies (eg, infliximab, adalimumab, golimumab) < 8 weeks prior to screening rectosigmoidoscopy.
  * Anti integrin antibodies (eg, vedolizumab) < 8 weeks prior to screening rectosigmoidoscopy.
  * IL 12/23 antagonist (eg, ustekinumab) < 8 weeks prior to screening rectosigmoidoscopy.
  * JAK inhibitors (eg, tofacitinib) < 4 weeks prior to screening rectosigmoidoscopy.
  * Any other commercially approved biologic agent or targeted small molecule < 8 weeks prior to screening rectosigmoidoscopy or < 5 half lives prior to screening rectosigmoidoscopy, whichever is longer
  * Immunomodulatory medications, including oral cyclosporine, intravenous cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, thalidomide < 4 weeks prior to screening rectosigmoidoscopy.
  * Any investigational biologic therapy within 8 weeks prior to screening rectosigmoidoscopy or < 5 half-lives prior to screening rectosigmoidoscopy, whichever is longer.
  * Has used apheresis (eg, Adacolumnâ apheresis) < 2 weeks prior to screening rectosigmoidoscopy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (200):
- United States (63):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Birmingham Digestive Health Research, LLC, Homewood, Alabama
  - Arizona Health Research, Mesa, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC, Phoenix, Arizona
  - Southern California Research Center, Coronado, California
  - United Medical Doctors, Los Alamitos, California
  - Biopharma Informatic Incorporated, Los Angeles, California
  - Gastrointestinal Biosciences Clinical Trials Limited Liability Company, Los Angeles, California
  - University of California Irvine, Orange, California
  - Santa Maria Gastroenterology Medical Group, Santa Maria, California
  - Clinical Trials Management Services LLC, Thousand Oaks, California
  - Gastroenterology Center of Connecticut, PC, Hamden, Connecticut
  - West Central Gastroenterology, Clearwater, Florida
  - Homestead Associates In Research Inc, Homestead, Florida
  - Indian Health Service Health Research, Kissimmee, Florida
  - Lake Center for Clinical Research, Lady Lake, Florida
  - Auzmer Research, Lakeland, Florida
  - University of Miami Hospital and Clinic, Miami, Florida
  - Ocala Gastrointestinal Research, LLC, Ocala, Florida
  - AdventHealth Medical Group Gastroenterology and Hepatology, Orlando, Florida
  - Infigo Clinical Research, Sanford, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Columbus Regional Research Institute, LLC, Columbus, Georgia
  - Grand Teton Research Group, Idaho Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Digestive Research Alliance of Michiana, South Bend, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mid-Atlantic GI Research, LLC, Greenbelt, Maryland
  - Harvard Medical School - Brigham and Womens Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, Troy, Michigan
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - Southern Therapy and Advanced Research LLC - Jackson, Jackson, Mississippi
  - Gastrointestinal Associates Research, LLC, Columbia, Missouri
  - Bvl Clinical Research, Liberty, Missouri
  - Interspond - Las Vegas Medical Research, Las Vegas, Nevada
  - Sanmora Bespoke Clinical Research Solutions, East Orange, New Jersey
  - Aga Clinical Research Associates LLC, Egg Harbor, New Jersey
  - Affiliates in Gastroenterology Digestive Disease Research, Florham Park, New Jersey
  - Atlantic Digestive Health Institute, Morristown, New Jersey
  - Premier Health Research LLC, Sparta, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - New York University Grossman School of Medicine and New York University Langone Hospitals, Lake Success, New York
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Digestive Specialists Inc Research, LLC, Springboro, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Guthrie Robert Packer Hospital, Sayre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Columbia Digestive Health Research LLC, Columbia, South Carolina
  - Wake Research-ClinSearch, LLC, Chattanooga, Tennessee
  - Digestive Health Research, LLC, Hermitage, Tennessee
  - Great Lakes Research Insititute El Paso Research, El Paso, Texas
  - Digestive Health Associates, Houston, Texas
  - Digestive Research of Central Texas, LLC, Waco, Texas
  - Digestive Health Research of North Texas LLC, Wichita Falls, Texas
  - Emeritas Research Group, Lansdowne Town Center, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - North Richmond Health Research, Richmond, Virginia
  - GI Select Health Research LLC, Richmond, Virginia
  - Hunter Holmes McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Argentina (6):
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Clinica Independencia, Munro, Buenos Aires
  - Cer Instituto Medico, Quilmes, Buenos Aires
  - CardioAlem Investigaciones, San Isidro, Buenos Aires
  - Hospital Privado Centro Medico de Cordoba SA, Córdoba, Córdoba Province
  - Fundacion Estudios Clinicos, Rosario, Santa Fe Province
- Austria (3):
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Landeskrankenhaus Salzburg, Salzburg
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
- Bulgaria (3):
  - Second Multiprofile Hospital for Active Treatment - Sofia EAD, Sofia
  - Diagnostic-Consultative Center Convex EOOD, Sofia
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment Mladost EOOD, Sofia
- Canada (3):
  - South Edmonton Gastroenterology, Edmonton, Alberta
  - London Health Sciences Centre, University Hospital, London, Ontario
  - TIDHI Innovation Incorporated, Toronto, Ontario
- Czechia (5):
  - Hepato-Gastroenterologie HK sro, Hradec Králové
  - Nemocnice Pardubickeho kraje as, Pardubicka nemocnice, Pardubice
  - Nemocnice Milosrdnych sester sv Karla Boromejskeho v Praze, Prague
  - Axon Clinical sro, Prague
  - Krajska zdravotni as - Masarykova nemocnice Usti nad Labem oz, Ústí nad Labem
- Denmark (4):
  - Aalborg Universitetshospital, Aalborg
  - Herlev Hospital, Herlev
  - Hvidovre Hospital, Hvidovre
  - Bispebjerg Hospital, København NV
- Helsinki University Central Hospital, Helsinki, Finland
- France (6):
  - Centre Hospitalier Universitaire Amiens Picardie, Amiens
  - Centre Hospitalier Universitaire de Montpellier - Hopital Saint Eloi, Montpellier
  - Centres Medicaux Chirurgicaux Ambroise Pare Hartmann, Neuilly-sur-Seine
  - Centre Hospitalier Universitaire Archet 2, Nice
  - Centre Hospitalier Universitaire Nord de Saint Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - Centre Hospitalier Universitaire de Nancy - Hôpital de Brabois, Vandœuvre-lès-Nancy
- Germany (6):
  - Gastro-Studien GbR Studienzentrum, Berlin
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Ulm, Ulm
- Greece (8):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - General Hospital Evangelismos, Athens
  - Laiko General Hospital of Athens, Athens
  - University Hospital Attikon, Haidari
  - Venizeleio General Hospital, Heraklion
  - University Hospital of Heraklion, Heraklion
  - University General Hospital of Ioannina, Ioannina
  - General University Hospital of Patras Panagia i Voithia, Pátrai
- Hungary (7):
  - Bekes Varmegyei Kozponti Korhaz Dr Rethy Pal Tagkorhaz, Békéscsaba
  - MIND Klinika Kft, Budapest
  - Clinexpert Kft, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Altalanos Orvostudomanyi Kar, Szeged
  - Clinfan Kft, Szekszárd
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz, Tatabánya
- Italy (8):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Universitaria Renato Dulbecco, Catanzaro
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino IRCCS, Genoa
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Ospedale Sacro Cuore Don Calabria, Negrar VR
  - Ospedale Sandro Pertini, Roma
- Japan (21):
  - Tsujinaka Hospital Kashiwanoha, Kashiwa-shi, Chiba
  - Toho University Sakura Medical Center, Sakura-shi, Chiba
  - Kitakyushu Municipal Medical Center, Kitakyushu-shi, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - Matsunami General Hospital, Hashima-gun, Gifu
  - Hakodate Central General Hospital, Hakodate-shi, Hokkaido
  - Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Aoyama Clinic GI Endoscopy and IBD Center, Kobe, Hyōgo
  - Gokeikai Ofuna Chuo Hospital, Kamakura-shi, Kanagawa
  - Takagi Clinic, Sendai, Miyagi
  - Miyazaki Prefectural Miyazaki Hospital, Miyazaki, Miyazaki
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Nara Medical University Hospital, Kashihara-shi, Nara
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Tokyo Medical and Dental University Hospital, Bunkyo-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - Kyorin University Hospital, Mitaka-shi, Tokyo
  - Ome Medical Center, Ome-shi, Tokyo
  - Medical Corporation ENEXT Ikebukuro West Gate Hospital, Toshima-ku, Tokyo
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Gastro Centrs, Riga
- Mexico (6):
  - Clinica de Investigacion en Reumatologia y Obesidad SC, Guadalajra, Jalisco
  - Investigacion Biomedica para el Desarrollo de Farmacos SA de CV, Zapopan, Jalisco
  - Clinicos Asociados BOCM SC, Mexico City, Mexico City
  - CRI Centro Regiomontano de Investigacion SC, Monterrey, Nuevo León
  - Hospital San Jose Tec Salud Fundacion Santos y de la Garza Evia IBP, Monterrey, Nuevo León
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada SC, Culiacán, Sinaloa
- Netherlands (3):
  - Leids Universitair Medisch Centrum, Leiden
  - Elisabeth TweeSteden Ziekenhuis, Tilburg
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (8):
  - NZOZ Twoje Zdrowie EL Spzoo, Elblag
  - Centrum Medyczne Med-Gastr Sp zoo, Lodz
  - Centrum Badawcze Panaceum Agnieszka Brzezicka Magdalena Lenkiewicz Spzoo, Malbork
  - Oleg Tyszkiwski Centrum Gastrologiczne Gorczyn Oleg Tyszkiwski, Poznan
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - BodyClinic spolka z ograniczona odpowiedzialnoscia, Warsaw
  - EuroMediCare Przychodnia Specjalistyczna we Wroclawiu, Wroclaw
  - Centrum Medyczne Melita Medical, Wroclaw-Krzyki
- Romania (6):
  - Spitalul Universitar de Urgenta Militar Central Dr Carol Davila, Bucharest
  - Clinica Medicum, Bucharest
  - Memorial Healthcare International SRL, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Pelican, Oradea
- Slovakia (3):
  - Fakultna Nemocnica s poliklinikou FD Roosevelta Banska Bystrica, Banská Bystrica
  - Endomed, sro, Košice
  - Gastro I, sro, Prešov
- South Korea (5):
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Wonju Severance Christian Hospital, Wonju-si, Gangwon-do
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
- Switzerland (4):
  - Inselspital Bern, Bern
  - Intesto BE, Bern
  - Kantonsspital St Gallen, Sankt Gallen
  - Universitaetsspital Zuerich, Zurich
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (9):
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Antalya Egitim ve Arastirma Hastanesi, Antalya
  - Uludag Universitesi Tip Fakultesi Hastanesi, Bursa
  - Gaziantep Universitesi Tip Fakultesi Hastanesi, Gaziantep
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Dokuz Eylul Universitesi Tip Fakultesi Hastanesi, Izmir
  - Kocaeli Universitesi Tip Fakultesi Hastanesi, Kocaeli
  - Mersin Universitesi Tip Fakultesi Hastanesi, Mersin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 200 centers in 26 countries (Argentina, Austria, Belgium, Bulgaria, Canada, Czech Republic, Denmark, Finland, France, Germany, Greece, Hungary, Italy, Japan, Latvia, Mexico, Netherlands, Poland, Romania, Slovakia, South Korea, Spain, Switzerland, Taiwan, Turkey, and the United States) between January 2022 to October 2024.
Pre-assignment Details: Participants were randomized to receive 1 of 3 efavaleukin alfa doses or placebo during a 12-week induction period in 1:1:1:1 ratio. Participants who completed the 12-week induction period had the option to enter an exploratory long-term treatment (LTT) period for up to 40 weeks (total of up to 52 weeks of treatment). The study was terminated due to meeting a predefined futility criterion and not related to any safety concerns.
Groups:
- Placebo Q2W: Participants received placebo matching efavaleukin alfa every 2 weeks (Q2W) through a subcutaneous (SC) injection for up to 52 weeks. Participants randomized to placebo who achieved clinical response continued in placebo, while those who did not achieve clinical response at week 12 were reassigned in a blinded manner to efavaleukin alfa 1100 micrograms (mcg) Q2W during the LTT period.
- Efavaleukin Alfa 400 µg Q2W: Participants received efavaleukin alfa 400 mcg Q2W through a SC injection for up to 52 weeks.
- Efavaleukin Alfa 1100 µg Q2W: Participants received efavaleukin alfa 1100 mcg Q2W through a SC injection for up to 52 weeks.
- Efavaleukin Alfa 1800 µg Q2W: Participants received efavaleukin alfa 1800 mcg Q2W through a SC injection for up to 52 weeks.
Period: Overall Study
Arm/Group | Placebo Q2W | Efavaleukin Alfa 400 µg Q2W | Efavaleukin Alfa 1100 µg Q2W | Efavaleukin Alfa 1800 µg Q2W
Started | 57 | 57 | 54 | 53
Responder at Week 12 in Placebo Q2W | 15 | 0 | 0 | 0
Non-responder at Week 12 in Placebo Q2W | 42 | 0 | 0 | 0
Completed (The completed milestone reflects the participants who entered the LTT period and completed the overall study.) | 10 | 14 | 14 | 6
Not Completed | 47 | 43 | 40 | 47
Not completed — Protocol-specified criteria | 2 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 34 | 30 | 29 | 35
Not completed — Decision by sponsor | 10 | 13 | 11 | 9
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants randomized.
Groups:
- Placebo Q2W: Participants received placebo matching efavaleukin alfa Q2W through a SC injection for up to 52 weeks. Participants randomized to placebo who achieved clinical response continued in placebo, while those who did not achieve clinical response at week 12 were reassigned in a blinded manner to efavaleukin alfa 1100 mcg Q2W during the LTT period.
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Efavaleukin Alfa 400 µg Q2W | Efavaleukin Alfa 1100 µg Q2W | Efavaleukin Alfa 1800 µg Q2W | Total
Number analyzed (Participants) | 57 | 57 | 54 | 53 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (14.8) | 43.8 (14.4) | 44.7 (16.8) | 44.6 (15.2) | 44.3 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 17 | 17 | 23 | 86
  Male | 28 | 40 | 37 | 30 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 8 | 5 | 30
  Not Hispanic or Latino | 42 | 47 | 45 | 42 | 176
  Unknown or Not Reported | 4 | 4 | 1 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 2
  Asian | 8 | 9 | 7 | 5 | 29
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 45 | 40 | 45 | 39 | 169
  Other | 0 | 3 | 1 | 2 | 6
  Missing | 4 | 4 | 0 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Remission at Week 12
Description: Clinical remission was defined as a modified Mayo score of 0 to 2, including a rectal bleeding subscore of 0, a stool frequency subscore of 0 or 1, and a centrally read endoscopy subscore of 0 or 1 (modified so that 1 did not include friability). The modified Mayo score was the total Mayo score ranged from 0 to 9 points, with higher scores indicating more severe disease.
Time Frame: Week 12
Population: FAS included all participants randomized. Only participants with available data were included in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Efavaleukin Alfa 400 µg Q2W | Efavaleukin Alfa 1100 µg Q2W | Efavaleukin Alfa 1800 µg Q2W
Number analyzed (Participants) | 53 | 51 | 52 | 48
percentage of participants | 7.5 | 9.8 | 9.6 | 10.4
Statistical Analysis 1: Comparison: Placebo Q2W vs Efavaleukin Alfa 400 µg Q2W; Test type: Superiority; p = 0.70, Logistic regression model — P-value was unadjusted and obtained from logistic regression model including stratification factors as covariates (prior experience with ≥1 biologic or targeted small molecule, corticosteroid use at randomization) using nonresponder imputation (NRI); Difference percentage (%) = 2.1, 95% CI 2-sided [-8.6 to 12.8]
Statistical Analysis 2: Comparison: Placebo Q2W vs Efavaleukin Alfa 1100 µg Q2W; Test type: Superiority; p = 0.72, Logistic regression model — P-value was unadjusted and obtained from logistic regression model including stratification factors as covariates (prior experience with ≥1 biologic or targeted small molecule, corticosteroid use at randomization) using NRI; Difference % = 2.0, 95% CI 2-sided [-8.6 to 12.6]
Statistical Analysis 3: Comparison: Placebo Q2W vs Efavaleukin Alfa 1800 µg Q2W; Test type: Superiority; p = 0.58, Logistic regression model — [p-value comment as in outcome 1, analysis 2]; Difference % = 3.1, 95% CI 2-sided [-8.0 to 14.2]

2. Secondary Outcome: Percentage of Participants With Clinical Response at Week 12
Description: Clinical response was defined as a decrease from baseline in the modified Mayo score of ≥ 2 points and at least a 30% reduction from baseline, and a decrease in the rectal bleeding subscore of ≥ 1 or an absolute rectal bleeding subscore of 0 or 1. The modified Mayo score was the total Mayo score without the physician's global assessment subscore and ranged from 0 to 9 points, with higher scores indicating more severe disease. Only participants who had the opportunity to complete the visit by the date of the decision for the study termination were included in this outcome measure. Efficacy data collected after this date were censored and excluded from analyses.
Time Frame: Baseline and Week 12
Population: FAS included all participants randomized. Only participants with available data were included in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Efavaleukin Alfa 400 µg Q2W | Efavaleukin Alfa 1100 µg Q2W | Efavaleukin Alfa 1800 µg Q2W
Number analyzed (Participants) | 53 | 51 | 52 | 48
percentage of participants | 20.8 | 19.6 | 25.0 | 25.0
Statistical Analysis 1: Comparison: Placebo Q2W vs Efavaleukin Alfa 400 µg Q2W; Test type: Superiority; p = 0.89, Logistic regression model — [p-value comment as in outcome 1, analysis 2]; Difference % = -1.1, 95% CI 2-sided [-16.3 to 14.2]
Statistical Analysis 2: Comparison: Placebo Q2W vs Efavaleukin Alfa 1100 µg Q2W; Test type: Superiority; p = 0.56, Logistic regression model — [p-value comment as in outcome 1, analysis 2]; Difference % = 4.7, 95% CI 2-sided [-11.1 to 20.6]
Statistical Analysis 3: Comparison: Placebo Q2W vs Efavaleukin Alfa 1800 µg Q2W; Test type: Superiority; p = 0.59, Logistic regression model — [p-value comment as in outcome 1, analysis 2]; Difference % = 4.5, 95% CI 2-sided [-11.7 to 20.7]

3. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Week 12
Description: Endoscopic remission was defined as a Mayo centrally read endoscopy subscore of 0 or 1 (modified so that a score of 1 did not include friability). The modified Mayo score was the total Mayo score ranged from 0 to 9 points, with higher scores indicating more severe disease.
Time Frame: Week 12
Population: FAS included all participants randomized. Only participants with available data were included in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Efavaleukin Alfa 400 µg Q2W | Efavaleukin Alfa 1100 µg Q2W | Efavaleukin Alfa 1800 µg Q2W
Number analyzed (Participants) | 53 | 51 | 52 | 48
percentage of participants | 11.3 | 15.7 | 11.5 | 12.5
Statistical Analysis 1: Comparison: Placebo Q2W vs Efavaleukin Alfa 400 µg Q2W; Test type: Superiority; p = 0.52, Logistic regression model — [p-value comment as in outcome 1, analysis 2]; Difference % = 4.2, 95% CI 2-sided [-8.7 to 17.2]
Statistical Analysis 2: Comparison: Placebo Q2W vs Efavaleukin Alfa 1100 µg Q2W; Test type: Superiority; p = 0.97, Logistic regression model — [p-value comment as in outcome 1, analysis 2]; Difference % = 0.2, 95% CI 2-sided [-11.8 to 12.2]
Statistical Analysis 3: Comparison: Placebo Q2W vs Efavaleukin Alfa 1800 µg Q2W; Test type: Superiority; p = 0.82, Logistic regression mode — [p-value comment as in outcome 1, analysis 2]; Difference % = 1.5, 95% CI 2-sided [-11.1 to 14.0]

4. Secondary Outcome: Percentage of Participants With Symptomatic Remission at Week 12
Description: Symptomatic remission was defined as Mayo stool frequency subscore of 0 or 1 and rectal bleeding subscore of 0. The modified Mayo score was the total Mayo score ranged from 0 to 9 points, with higher scores indicating more severe disease.
Time Frame: Week 12
Population: FAS included all participants randomized. Only participants with available data were included in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Efavaleukin Alfa 400 µg Q2W | Efavaleukin Alfa 1100 µg Q2W | Efavaleukin Alfa 1800 µg Q2W
Number analyzed (Participants) | 53 | 51 | 52 | 48
percentage of participants | 15.1 | 17.6 | 23.1 | 22.9
Statistical Analysis 1: Comparison: Placebo Q2W vs Efavaleukin Alfa 400 µg Q2W; Test type: Superiority; p = 0.72, Logistic regression model — [p-value comment as in outcome 1, analysis 2]; Difference % = 2.6, 95% CI 2-sided [-11.6 to 16.7]
Statistical Analysis 2: Comparison: Placebo Q2W vs Efavaleukin Alfa 1100 µg Q2W; Test type: Superiority; p = 0.28, Logistic regression model — [p-value comment as in outcome 1, analysis 2]; Difference % = 8.3, 95% CI 2-sided [-6.6 to 23.1]
Statistical Analysis 3: Comparison: Placebo Q2W vs Efavaleukin Alfa 1800 µg Q2W; Test type: Superiority; p = 0.30, Logistic regression model — [p-value comment as in outcome 1, analysis 2]; Difference % = 8.1, 95% CI 2-sided [-7.1 to 23.3]

5. Secondary Outcome: Percentage of Participants With Combined Endoscopic Remission and Histologic Remission of the Colon Tissue at Week 12
Description: Combined endoscopic and histologic remission was defined as combined endoscopic remission (Mayo centrally read endoscopy subscore of 0 or 1) and histologic remission of the colon tissue (Geboes Score < 2.0; no neutrophils in epithelium crypts or lamina propria and no increase in eosinophils, no crypt destruction and no erosions, ulcerations or granulation tissue). Geobes score was defined as: grade 0, structural (architectural change); grade 1, chronic inflammatory infiltrate; grade 2A, lamina propria eosinophils; grade 2B, lamina propria neutrophils; grade 3, neutrophils in epithelium; grade 4, crypt destruction; and grade 5, erosion or ulceration. Each grade included subscores that indicated degree of abnormality, with subscores of 0 indicating normal appearance and higher subscores indicating increasingly abnormal appearance. The modified Mayo score was total Mayo score ranged from 0 to 9 points, with higher scores indicating more severe disease.
Time Frame: Week 12
Population: FAS included all participants randomized. Only participants with available data were included in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Efavaleukin Alfa 400 µg Q2W | Efavaleukin Alfa 1100 µg Q2W | Efavaleukin Alfa 1800 µg Q2W
Number analyzed (Participants) | 53 | 51 | 52 | 48
percentage of participants | 0.0 | 7.8 | 1.9 | 0.0
Statistical Analysis 1: Comparison: Placebo Q2W vs Efavaleukin Alfa 400 µg Q2W; Test type: Superiority; p = 0.11, Logistic regression model — [p-value comment as in outcome 1, analysis 2]; Difference % = 8.46, 95% CI 2-sided [0.0 to 16.9]
Statistical Analysis 2: Comparison: Placebo Q2W vs Efavaleukin Alfa 1100 µg Q2W; Test type: Superiority; p = 0.46, Logistic regression model — [p-value comment as in outcome 1, analysis 2]; Difference % = 2.18, 95% CI 2-sided [-3.4 to 7.7]
Statistical Analysis 3: Comparison: Placebo Q2W vs Efavaleukin Alfa 1800 µg Q2W; Test type: Superiority; p = 0.94, Logistic regression model — [p-value comment as in outcome 1, analysis 2]; Difference % = 0.14, 95% CI 2-sided [-4.0 to 4.3]

6. Secondary Outcome: Change From Baseline in Histological Score at Week 12 as Measured by the Geboes Score
Description: The Geboes score was an instrument used to standardize histologic assessment in ulcerative colitis (UC). It comprised seven categories (or grades), each describing a histologic feature. These categories were as follows: grade 0, structural (architectural change); grade 1, chronic inflammatory infiltrate; grade 2A, lamina propria eosinophils; grade 2B, lamina propria neutrophils; grade 3, neutrophils in epithelium; grade 4, crypt destruction; and grade 5, erosion or ulceration. Each grade included subscores that indicated the degree of abnormality observed for that histologic feature. Subscores ranged from 0 to 5.4, where a score of 0 indicated no or minimal inflammation, and a maximum score of 5.4 reflected severe histological activity.
Time Frame: Baseline to Week 12
Population: FAS included all participants randomized. Only participants with available data were included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo Q2W | Efavaleukin Alfa 400 µg Q2W | Efavaleukin Alfa 1100 µg Q2W | Efavaleukin Alfa 1800 µg Q2W
Number analyzed (Participants) | 51 | 51 | 49 | 46
score on scale | -0.53 (1.31) | -0.30 (1.39) | -0.34 (1.49) | -0.45 (1.04)
Statistical Analysis 1: Comparison: Placebo Q2W vs Efavaleukin Alfa 400 µg Q2W; Test type: Superiority; p = 0.39, ANCOVA — P-value was obtained from the analysis of covariance (ANCOVA) model which includes stratification factors (prior experience with ≥ 1 biologic or targeted small molecule, corticosteroid use at randomization) as covariates; Treatment Difference = 0.2, 95% CI 2-sided [-0.3 to 0.7]
Statistical Analysis 2: Comparison: Placebo Q2W vs Efavaleukin Alfa 1100 µg Q2W; Test type: Superiority; p = 0.49, ANCOVA — P-value was obtained from the ANCOVA model which includes stratification factors (prior experience with ≥ 1 biologic or targeted small molecule, corticosteroid use at randomization) as covariates; Treatment Difference = 0.2, 95% CI 2-sided [-0.3 to 0.7]
Statistical Analysis 3: Comparison: Placebo Q2W vs Efavaleukin Alfa 1800 µg Q2W; Test type: Superiority; p = 0.76, ANCOVA — [p-value comment as in outcome 6, analysis 2]; Treatment Difference = 0.1, 95% CI 2-sided [-0.5 to 0.6]

7. Secondary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were events categorized as adverse events (AEs) that started on or after the first dose of investigational product (IP), and up to 12 weeks in induction period.
Time Frame: Up to 12 weeks
Population: Safety analysis set included all participants randomized and received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | Efavaleukin Alfa 400 µg Q2W | Efavaleukin Alfa 1100 µg Q2W | Efavaleukin Alfa 1800 µg Q2W
Number analyzed (Participants) | 57 | 57 | 53 | 53
Participants | 33 | 42 | 42 | 46

ADVERSE EVENTS:
Time Frame: All-cause mortality: From enrollment until the end of study (EOS); median (min, max) time on study was 22.49 (2.85, 83.14) weeks. Serious AEs and other AEs: From first dose of study drug until the EOS; median (min, max) duration was 22.49 (2.85, 83.14) weeks.
Description: All-cause mortality is reported for all randomized participants; serious and other AEs are reported for all participants who received at least one dose of study drug. One participant who was a Week 12 responder was excluded from the Placebo Q2W in the LTT, and did not receive placebo in the LTT.
Groups:
- Placebo Q2W in Induction: Participants were randomized to receive placebo matching efavaleukin alfa once Q2W through a SC injection in the induction period (from Weeks 1 to 12).
- Placebo Q2W in LTT: Participants randomized to placebo Q2W during the induction period (from Weeks 1 to 12) who achieved a clinical response at Week 12 and continued to receive placebo Q2W throughout the LTT period (from Weeks 13 to 52).
- Efavaleukin Alfa 1100 µg Q2W LTT: Participants randomized to placebo Q2W during the induction period (from Weeks 1 to 12) who did not achieve a clinical response at Week 12 and received efavaleukin alfa 1100 mcg administered Q2W through a SC injection throughout the LTT period (from Weeks 13 to 52).
Arm/Group | Placebo Q2W in Induction | Placebo Q2W in LTT | Efavaleukin Alfa 1100 µg Q2W LTT | Efavaleukin Alfa 400 µg Q2W | Efavaleukin Alfa 1100 µg Q2W | Efavaleukin Alfa 1800 µg Q2W
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/14 | 0/42 | 0/57 | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 5/57 | 0/14 | 5/42 | 3/57 | 7/53 | 9/53
Other Adverse Events (participants affected / at risk) | 39/57 | 9/14 | 29/42 | 47/57 | 44/53 | 46/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W in Induction (N=57) | Placebo Q2W in LTT (N=14) | Efavaleukin Alfa 1100 µg Q2W LTT (N=42) | Efavaleukin Alfa 400 µg Q2W (N=57) | Efavaleukin Alfa 1100 µg Q2W (N=53) | Efavaleukin Alfa 1800 µg Q2W (N=53)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 4 | 0 | 4 | 2 | 4 | 5
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W in Induction (N=57) | Placebo Q2W in LTT (N=14) | Efavaleukin Alfa 1100 µg Q2W LTT (N=42) | Efavaleukin Alfa 400 µg Q2W (N=57) | Efavaleukin Alfa 1100 µg Q2W (N=53) | Efavaleukin Alfa 1800 µg Q2W (N=53)
Anaemia (Blood and lymphatic system disorders) | 6 | 0 | 6 | 4 | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 1 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 2 | 4 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 4 | 0
Colitis ulcerative (Gastrointestinal disorders) | 14 | 4 | 9 | 12 | 9 | 5
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 3 | 3
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 1 | 5
Asthenia (General disorders) | 1 | 0 | 1 | 1 | 3 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 3
Fatigue (General disorders) | 2 | 0 | 2 | 2 | 4 | 8
Influenza like illness (General disorders) | 1 | 0 | 1 | 1 | 4 | 0
Injection site erythema (General disorders) | 11 | 0 | 10 | 24 | 22 | 30
Injection site oedema (General disorders) | 0 | 0 | 0 | 2 | 3 | 3
Injection site pain (General disorders) | 3 | 0 | 3 | 2 | 3 | 4
Injection site pruritus (General disorders) | 3 | 0 | 2 | 12 | 8 | 11
Injection site rash (General disorders) | 1 | 0 | 1 | 3 | 4 | 4
Injection site reaction (General disorders) | 3 | 0 | 3 | 4 | 3 | 6
Injection site swelling (General disorders) | 3 | 0 | 2 | 9 | 6 | 9
Pyrexia (General disorders) | 2 | 0 | 2 | 9 | 9 | 5
COVID-19 (Infections and infestations) | 2 | 1 | 1 | 2 | 1 | 3
Influenza (Infections and infestations) | 4 | 1 | 3 | 1 | 0 | 3
Nasopharyngitis (Infections and infestations) | 3 | 0 | 3 | 3 | 4 | 2
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 0 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 2 | 3 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 4 | 9 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 3 | 1
Headache (Nervous system disorders) | 3 | 1 | 2 | 5 | 5 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 7 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 3 | 7
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 3 | 1 | 7 | 10
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 1
Oral hyperaesthesia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 1
Varicose vein (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to meeting a predefined futility criterion and not related to any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT04987307/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT04987307/SAP_001.pdf